CLINICAL TRIAL: NCT03000946
Title: Prevention of Postoperative Pancreatic Fistula by SOMATOSTATIN Compared to OCTREOTIDE: Prospective, Randomized, Controlled Study
Brief Title: Prevention of Postoperative Pancreatic Fistula by Somatostatin
Acronym: PREFIPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P150915; 2016-001673-32 (EudraCT Number)
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Surgery
Keywords: Pancreatectomy; Somatostatin analogue; Octreotide; Pancreatic fistula
MeSH Terms: conditions — Pancreatic Fistula | interventions — Somatostatin; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Somatostatin (Experimental): Continuous intravenous infusion of somatostatin-14, 6 mg per day during 6.5 days
  Interventions: Drug: Somatostatin
- Octreotide (Active Comparator): Subcutaneous octreotide 100 μg 3 times a day for 6.5 days.
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Somatostatin — Lyophilisate and solution for IV use (glass ampoule of lyophilisate + 1 ml glass ampoule of solvent) 6 mg per day Continuous intravenous infusion for 6,5 days
  Other Names: Somatostatine Eumedica
  Arms: Somatostatin
Drug: Octreotide — Solution for Subcutaneous use 100μg, every 8 hours Subcutaneous injection for 6,5 days
  Other Names: Siroctid
  Arms: Octreotide

SUMMARY:
The purpose of this study is to determine whether somatostatin is more effective that octreotide in the prevention of post-pancreatectomy pancreatic fistula

DETAILED DESCRIPTION:
Prevention of pancreatic fistula remains a major challenge for surgeons, and various technical and pharmacological intervention have been investigated, with conflicting results.

Despite several prospective studies, and metaanalyses, the prophylactic role on pancreatic fistula of octreotide, remains controversial, even if recommended for routine use in patients undergoing pancreatic resection.

In view of recent result, the investigators can hypothesize that higher affinity for somatostatin-receptor lead to stronger pancreatic exocrine secretion inhibition, and better pancreatic fistula prevention.

Consequently, continuous intravenous infusion of somatostatin-14, the natural peptide hormone, associated with 10 to 50 time stronger affinity with all somatostatin receptor, will be associated with a improved pancreatic fistula prevention compared to octreotide.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years or greater
* Signed informed consent
* Candidate for pancreaticoduodenectomy or distal pancreatectomy with or without splenectomy

Exclusion Criteria:

* Patient with radiation therapy
* Patient with neoadjuvant chemotherapy within 4 weeks before surgery
* Pregnancy
* Breastfeeding
* Patients who have any current or prior medical condition that may interfere with the conduct of the study or the evaluation of its results in the opinion of the Investigator
* Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to inclusion
* Known hypersensitivity to somatostatin or somatostatin analogues or any component of the somatostatin or octreotide long-acting release (LAR) or s.c. formulations
* Patient previously treated with somatostatin or somatostatin analogues or any component of the somatostatin or octreotide LAR or s.c. formulations
* Patients treated by ciclosporin
* Patient without health insurance or social security
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
≥ grade B or C postoperative pancreatic fistula as defined by the International Study Group of Pancreatic Fistula (ISGPF) classification | 90 days

SECONDARY OUTCOMES:
≥grade 3 pancreatic complication rates (fistula, leak, and abscess) | 60 days
  as defined by the MSKCC surgical secondary events system
Overall pancreatic fistula rate (grade A,B and C) | 90 days
  previous ISGPF classification
Overall pancreatic fistula rate (grade B and C) | 90 days
  last ISGPF classification
Overall complication rate (grade 1 to 5) | 90 days
  according to Clavien-Dindo classification
Severe complication rate (grade 3 to 5) | 90 days
  according to Clavien-Dindo classification
Mortality (grade 5) | 90 days
  according to Clavien-Dindo classification
Overall duration of drainage | 90 days
  required in patients who develop pancreatic complications (date pancreatic complication identified - date drain removed)
Overall length of stay | 90 days
Re-admission rate | 90 days
Cost effectiveness | 90 days
Fistula according to possible new definition of the ISGPF group | 90 days
Postoperative quality of life after pancreatic surgery | 7 days after surgery
  only in patients undergoing pancreaticoduodenectomy

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien GAUJOUX, MD, PhD, Principal Investigator — La Pitié Salpêtrière Hospital, AP-HP; Bertrand DOUSSET, MD, PhD, Study Chair — Cochin Hospital, AP-HP
Locations (2):
- France (2):
  - Cochin Hospital, Paris, Paris
  - La Pitié Salpêtrière Hospital, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaujoux S, Regimbeau JM, Piessen G, Truant S, Foissac F, Barbier L, Buc E, Adham M, Fuks D, Deguelte S, Muscari F, Sulpice L, Vaillant JC, Schwarz L, Sa Cunha A, Muzzolini M, Dousset B, Sauvanet A; Collaborators. Somatostatin Versus Octreotide for Prevention of Postoperative Pancreatic Fistula: The PREFIPS Randomized Clinical Trial: A FRENCH 007-ACHBT Study. Ann Surg. 2024 Aug 1;280(2):179-187. doi: 10.1097/SLA.0000000000006313. Epub 2024 Apr 25. PMID 38662619